CLINICAL TRIAL: NCT02092233
Title: A Two Arm, Multi-Site Clinical Evaluation of the ARIES HSV 1&2 Assay in Symptomatic Patients
Status: Completed | Type: Observational
Sponsor: Luminex Corporation (Industry)
Responsible Party: Sponsor
Organization: Luminex Molecular Diagnostics (Industry)
Other Study IDs: LMA-HSV-01-CS-001
Record Dates: First submitted 2014-03-17; First posted 2014-03-20 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2014-03

CONDITIONS: Herpes
Keywords: ARIES HSV 1&2
MeSH Terms: conditions — Herpes Simplex

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patient lesion swab specimens
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Blinded, Prospective Arm: The diagnostic accuracy for lesions from individuals suspected of having a herpes infection will be evaluated in prospectively collected, left-over de-identified, clinical specimens accrued between pre-defined dates.
- Blinded, Pre-selected Arm: For specimen types that are less common, banked, pre-selected, positive clinical specimens will be tested.

SUMMARY:
The ARIES HSV 1&2 Assay is a PCR based test for the direct detection and typing of herpes simplex virus (HSV 1 & 2) DNA.

The objective is to establish the diagnostic accuracy of ARIES HSV-1&2 Assay.

DETAILED DESCRIPTION:
The ARIES HSV 1&2 Assay is a polymerase chain reaction (PCR) based qualitative in vitro diagnostic test for the direct detection and typing of herpes simplex virus (HSV 1 & 2) DNA in male external and internal anogenital, female external and internal anogenital (vaginal), oral and skin lesion specimens.

The objective is to establish the diagnostic accuracy of ARIES HSV-1&2 Assay through a multi-site, method comparison on prospectively collected, left-over de-identified, clinical specimens (i.e. all-comers accrued at enrolled clinical sites between pre-determined dates) as an aid in the diagnosis of herpes infection.

ELIGIBILITY:
Inclusion Criteria:

The specimen is from one of the following lesion sources: male internal and external anogenital, female internal anogenital, female external anogenital, oral or skin The specimen is collected and maintained in unexpired Copan universal transport medium

Exclusion Criteria:

The specimen was not properly collected, transported or stored according to instructions provided by Sponsor

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Clinical lesions from pediatic or adult patients suspected of having herpes infection
Sampling Method: Probability Sample
Enrollment: 1963 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy will be expressed in terms of clinical sensitivity (or positive agreement) and specificity (or negative agreement). | Within the first year of sample collection

CONTACTS AND LOCATIONS:
Overall Officials: David Himsworth, Study Director — Luminex Corporation
Locations (3):
- United States (3):
  - Baystate Medical Center, Springfield, Massachusetts
  - Tricore, Albuquerque, New Mexico
  - Labcorp, Burlington, North Carolina